CLINICAL TRIAL: NCT06072963
Title: Combination of Intranasal Insulin With Oral Semaglutide to Improve Cognition and Cerebral Blood Flow: a Feasibility Study
Brief Title: COMMETS- Combination MCI Metabolic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Michal Schnaider Beeri, Ph.D., Director, Alzheimer's Research Center., Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2023001136
Record Dates: First submitted 2022-11-03; First posted 2023-10-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Metabolic Syndrome
Keywords: Alzheimer disease; Mild Cognitive Impairment; Metabolic syndrome; Dementia; Semaglutide; Intranasal insulin
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Metabolic Syndrome; Dementia | interventions — semaglutide; Insulin

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized with equal probability to each of the four study groups. Following the baseline assessment, participants will be assigned to one of the four intervention groups, as determined by an automated randomization algorithm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group 1 (Experimental): Will receive intranasal insulin therapy as well as Oral Semaglutide.
  Interventions: Drug: Semaglutide; Drug: Intranasal insulin
- Group 2 (Sham Comparator): Will receive active intranasal insulin therapy and placebo Oral Semaglutide.
  Interventions: Drug: Intranasal insulin; Other: Semaglutide placebo
- Group 3 (Sham Comparator): Will receive intranasal insulin placebo and active Oral Semaglutide .
  Interventions: Drug: Semaglutide; Other: Intranasal insulin placebo
- Group 4 (Placebo Comparator): Will receive intranasal insulin placebo and Oral Semaglutide placebo.
  Interventions: Other: Semaglutide placebo; Other: Intranasal insulin placebo

INTERVENTIONS:
Drug: Semaglutide — The medication is available in 3, 7, and 14-mg tablets for oral use. Participants will be instructed to start with an initiating dose of 3 mg once daily. If they do not experience adverse events (nausea, vomiting, and abdominal pain) then the dose will be titrated to 7 mg once daily after 30 days. Again, if the participant does not experience adverse events, the dose will be further titrated after 30 days to 14 mg once daily. This does will continue until the end of the study, at 12 months.
  Other Names: Rybelsus
  Arms: Group 1; Group 3
Drug: Intranasal insulin — The study will use the ViaNase; Kurve Technology intranasal device to administer insulin intra-nasally. This device has been used in other studies of persons with AD and has shown insulin penetration into the brain via CSF studies. Through sniffing, the medication crosses the blood-brain barrier (BBB) at the top of the nasal cavity. Participants will be instructed to press a switch that will turn on the device, engaging a pump that releases a nebulized stream of insulin through a nose piece into a nostril for 20 seconds (the device includes an electronic timer), after which the device switches off. The process is then repeated in the other nostril. The investigators decided on administration of 20IU of INI twice per day as the literature suggests this as the optimal dosage.
  Other Names: Actrapid
  Arms: Group 1; Group 2
Other: Semaglutide placebo — Rybelsus semaglutide - this medicine will simulate taking the pill Rybelsus /semaglutide once a day. A pill identical to the medicine pill will be given.
  Arms: Group 2; Group 4
Other: Intranasal insulin placebo — The placebo used in this study is saline. The investigators will administer saline, with exactly the same methods as the INI insulin (twice per day, 20 seconds each sniff, in each nostril.
  Arms: Group 3; Group 4

SUMMARY:
The investigators propose a proof of concept RCT (randomized clinical trial), testing the efficacy of intranasal insulin (INI) with semaglutide, a combination therapy with strong biological plausibility to benefit impaired cognition through vascular mechanisms, in older adults with MetS (metabolic syndrome) and MCI (Mild Cognitive Impairment), who are enriched for cerebrovascular disease and at high dementia risk. The study will focus on cognitive and biological outcomes, allowing identification of relevant mechanisms.

DETAILED DESCRIPTION:
The Specific Aims of the study are:

Aim 1. To examine the ease and precision of use of the intranasal device and once daily semaglutide pill.

Aim 2. To examine the adherence to the two types of treatment.

Aim 3. To examine the safety profile of the combination of intranasal insulin with semaglutide. The safety profile of each has been published broadly, but the safety of their combination has not been examined.

Aim 4. Although the primary goal of the pilot study is proof of concept essential to design a large combination therapy RCT, The investigators will compare the combination of intranasal insulin and semaglutide with the other three groups on a) cognition, b) cerebral blood flow (via ASL MRI), c) glucose uptake (via FDG PET), ADRD(Alzheimer's disease and related disorders)-related blood biomarkers (Aβ42/Aβ40 ratio, pTau181 and 231, NfL and GFAP), and expression of insulin signaling genes from brain derived exosomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MCI (based on a MOCA <27 and a clinical dementia rating scale [CDR] score of 0.5 representing questionable dementia).
* Diagnosis of MetS -requiring a) abdominal obesity (waist circumference >102cm for men and >88cm for women), and b) glucose intolerance (fasting glucose>110 mg/dL) and at least one of the following-c) dyslipidemia (high triglycerides [>150 mg/dL] and low HDL [<40mg/dL for men and <50 mg/dL for women]), or d) elevated blood pressure (>130/>85 mmHg).
* Fluent in Hebrew
* The study requires an active study partner

Exclusion Criteria:

* Diabetes (of any type)
* Taking medications that may affect glucose metabolism (including a GLP-1RA).
* Diagnosis of dementia and its subtypes, conditions that may directly affect cognition,
* short life expectancy or a medical condition that precludes consistent participation in the study,
* contraindications to either insulin or Semaglutide.
* Medications that may affect glucose metabolism such as corticosteroids.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive change - The effect of the combination of Semaglutide and intranasal insulin on cognitive functioning. | 12 months
  The cognitive outcome is a balanced composite sum of z-scores of four executive function tests (Trails B, Digit-Symbol, and Category Fluency (animals, fruits and vegetables), four episodic memory tests (immediate and delayed recall of the word list from the ADAS-Cog, and immediate and delayed recall of Logical Memory Story I from the Wechsler Memory Test). Z-scores are reversed if necessary so that a positive value refers to good cognition. Cognitive functioning will be measured at baseline, 6 months, and 12 months follow-ups.
Neuroimaging outcome -- The effect of the combination of Semaglutide and intranasal insulin on cerebral blood flow (CBF). | 6 months
  Change in CBF will be measured using Arterial Spin Labeling (ASL) brain magnetic resonance imaging (MRI) scans. The unit of cerebral blood flow from ASL is ml/100g/min, which means the amount of blood flow into 100g of tissue in one minute. Scans will be taken at baseline and 6 months follow-up. Baseline and 6 months scans will be compared and analyzed to assess change in blood flow between the time points.
Neuroimaging outcome -- The effect of the combination of Semaglutide and intranasal insulin on brain glucose intake. | 6 months
  Brain Glucose intake will be measured by [F18]FDG-PET: Voxel-wise standardized uptake value ratio (SUVR) images will be created in native MRI space with the pons as reference region. [F18]FDG values will be extracted from ADRD-vulnerable regions of interest (dorsolateral prefrontal cortex, medial and lateral temporal lobe, and medial and lateral parietal cortex). Scans will be taken at baseline and 6 months follow-up. Baseline and 6 months scans will be compared and analyzed to assess change in glucose intake between the time points.

SECONDARY OUTCOMES:
Change in specific cognitive domains - The effect of the combination of Semaglutide and intranasal insulin on executive functions and episodic memory. | 12 months
  Cognitive outcomes will be the domain-specific composites, for executive functions and episodic memory, by using four executive function tests (Trails B, Digit-Symbol, and Category Fluency [animals, fruits and vegetables), and four episodic memory tests (immediate and delayed recall of the word list from the ADAS-Cog, and immediate and delayed recall of Logical Memory Story I from the Wechsler Memory Test). Cognitive outcomes will be measured at baseline, 6 months, and 12 months follow-ups
Neuroimaging outcomes- The effect of the combination of Semaglutide and intranasal insulin on microstructural alterations indicative of tissue injury. | 6 months
  Changes in White matter hyperintensity (WMH) volume: Total WMH volume of presumed ischemic origin will be quantified from 3D T2-FLAIR brain MRI using the Lesion Segmentation Tool. T1-weighted volumetric scans will be used to derive intracranial volume. Scans will be taken at baseline and 6 months follow-up. Baseline and 6 months scans will be compared and analyzed to assess change in WMH volume between the time points.
Neuroimaging outcomes- The effect of the combination of Semaglutide and intranasal insulin on gray matter and hippocampal volume. | 6 months
  Changes in gray matter (GM) and hippocampal volumes: neurodegeneration will be measured using T1-weighted scans brain MRI scans. Regional cortical GM and hippocampal volumes will be extracted using FreeSurfer 7.1.1. and FSL. Scans will be taken at baseline and 6 months follow-up. Baseline and 6 months scans will be compared and analyzed to assess change in GM and hippocampal volumes between the time points.
Functional outcome - The effect of the combination of Semaglutide and intranasal insulin on functional performance. | 12 months
  Change in functional performance will be measured by the Clinical Dementia Rating (CDR) Scale Sum of Boxes (SB). The CDR-SB summarizes cognitive impairment in 6 domains (memory, orientation, judgment/problem-solving, community affairs, home/hobbies, and personal care) based on subject and informant interviews. Possible scores on the CDR are 0 (no impairment), 0.5 (very mild), 1 (mild), 2 (moderate), and 3 (severe). A maximal CDR-SB score is -18. CDR will be measured at baseline, 6 months, and 12 months follow-ups.
Functional outcome - The effect of the combination of Semaglutide with intranasal inulin on change in functional performance as measured by IADL (instrumental activities of daily living) questionnaires. | 12 months
  Functional Activities will be based on subject and informant interviews. Both ADLs (activities of daily living) and IADLs (instrumental ADLs) refer to key life tasks that need to be accomplish daily. ADLs, are more basic tasks that are essential to independent living. IADLs, are more complex tasks that are still a necessary part of everyday life. The study subjects are MCI, so mostly independent in ADLs. Therefore, the IADL questionnaire used in the "ADCS Prevention Instrument Project" will be used.
  IADL will be assessed at baseline, 6 months and 12 months. The range score is 0-45; a higher score means that the subject is more independent.
Functional outcome - The effect of the combination of Semaglutide and intranasal insulin on physical capacity | 6 months
  Physical capacity (PC) assessment (aerobic, balance, strength) includes grip strength, 6-m walk (6MWT), timed up and go (TUG), Berg balance testing (BBS), 30 Seconds Sit To Stand Test (STS), Four Square Step Test (FSST) and the Fried frailty scale. Based on the collected data, individuals will be categorized and assigned to 1 of 3 categories: low PC (LPC), medium PC (MPC), or normal PC (NPC). Participants will receive an LPC score if either standardized 6MWT/STS/Grip score is ≤ -2 standard deviation or BBS score ≤36 or TUG score between 21-30 or FSST score > 15 seconds or deemed as frail assessed by the Fried scale. Participants will have an MPC score if either the standardized 6MWT/STS/Grip score is between -2 and -1.5 or BBS score is between 37-45 or the TUG score is between 15-20 or FSST score is between 10.14-14.59 or determined as pre-frail by Fried scale. All other participants will be categorized as NPC. Physical capacity will be measured at baseline and 6 months follow-up.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers- Aβ. | 6 Months
  A lower amyloid beta (Aβ) 42/Aβ 40 ratio in plasma is associated with a higher risk of dementia. Aβ 42/Aβ 40 plasma ratio will be measured at baseline and 6 months followup and will be compared to assess change in ADRD-blood biomarkers between the time points.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers- P-tau181. | 6 Months
  A higher rate of P-tau181 in plasma is associated with a higher risk of dementia. Change in rate of plasma tau proteins in blood plasma from baseline to 6 months will be assessed.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers-P-tau231. | 6 Months
  A higher rate of P-tau231associated with a higher risk of dementia. Change in rate of plasma P-tau231 proteins from baseline to 6 months will be examined.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers- T-tau. | 6 Months
  A higher rate of T-tau associated with a higher risk of dementia. Change in rate of plasma T-tau proteins in blood plasma from baseline to 6 months will be examined.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers- Neurofilament light (NfL). | 6 Months
  A higher rate of neurofilament light (NfL) is associated with a higher risk of dementia. Change in rate of plasma tau proteins in blood plasma from baseline to 6 months will be examined.
Neurobiological outcome - The effect of the combination of Semaglutide and intranasal insulin on ADRD-blood biomarkers- glial fibrillary acidic protein (GFAP). | 6 Months
  A higher rate of glial fibrillary acidic protein (GFAP) is associated with a higher risk of dementia. Change in rate of plasma GFAP in blood plasma from baseline to 6 months will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Tal Davidy, Study Director — Sheba Medical Center; Michal Schnaider beeri, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Joseph Sagol Neuroscience center, Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Love S, Miners JS. Cerebrovascular disease in ageing and Alzheimer's disease. Acta Neuropathol. 2016 May;131(5):645-58. doi: 10.1007/s00401-015-1522-0. Epub 2015 Dec 28. PMID 26711459
- [Background] Daulatzai MA. Cerebral hypoperfusion and glucose hypometabolism: Key pathophysiological modulators promote neurodegeneration, cognitive impairment, and Alzheimer's disease. J Neurosci Res. 2017 Apr;95(4):943-972. doi: 10.1002/jnr.23777. Epub 2016 Jun 27. PMID 27350397
- [Background] Kim HW, Hong J, Jeon JC. Cerebral Small Vessel Disease and Alzheimer's Disease: A Review. Front Neurol. 2020 Aug 25;11:927. doi: 10.3389/fneur.2020.00927. eCollection 2020. PMID 32982937
- [Background] Gerstein HC, Colhoun HM, Dagenais GR, Diaz R, Lakshmanan M, Pais P, Probstfield J, Riesmeyer JS, Riddle MC, Ryden L, Xavier D, Atisso CM, Dyal L, Hall S, Rao-Melacini P, Wong G, Avezum A, Basile J, Chung N, Conget I, Cushman WC, Franek E, Hancu N, Hanefeld M, Holt S, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Cardona Munoz EG, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T; REWIND Investigators. Dulaglutide and cardiovascular outcomes in type 2 diabetes (REWIND): a double-blind, randomised placebo-controlled trial. Lancet. 2019 Jul 13;394(10193):121-130. doi: 10.1016/S0140-6736(19)31149-3. Epub 2019 Jun 9. PMID 31189511
- [Background] Gerstein HC, Hart R, Colhoun HM, Diaz R, Lakshmanan M, Botros FT, Probstfield J, Riddle MC, Ryden L, Atisso CM, Dyal L, Hall S, Avezum A, Basile J, Conget I, Cushman WC, Hancu N, Hanefeld M, Jansky P, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Munoz EGC, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T. The effect of dulaglutide on stroke: an exploratory analysis of the REWIND trial. Lancet Diabetes Endocrinol. 2020 Feb;8(2):106-114. doi: 10.1016/S2213-8587(19)30423-1. Epub 2020 Jan 7. PMID 31924562
- [Background] Cukierman-Yaffe T, Gerstein HC, Colhoun HM, Diaz R, Garcia-Perez LE, Lakshmanan M, Bethel A, Xavier D, Probstfield J, Riddle MC, Ryden L, Atisso CM, Hall S, Rao-Melacini P, Basile J, Cushman WC, Franek E, Keltai M, Lanas F, Leiter LA, Lopez-Jaramillo P, Pirags V, Pogosova N, Raubenheimer PJ, Shaw JE, Sheu WH, Temelkova-Kurktschiev T. Effect of dulaglutide on cognitive impairment in type 2 diabetes: an exploratory analysis of the REWIND trial. Lancet Neurol. 2020 Jul;19(7):582-590. doi: 10.1016/S1474-4422(20)30173-3. PMID 32562683
- [Background] Wu JH, Haan MN, Liang J, Ghosh D, Gonzalez HM, Herman WH. Impact of antidiabetic medications on physical and cognitive functioning of older Mexican Americans with diabetes mellitus: a population-based cohort study. Ann Epidemiol. 2003 May;13(5):369-76. doi: 10.1016/s1047-2797(02)00464-7. PMID 12821276
- [Background] Chen Y, Zhou K, Wang R, Liu Y, Kwak YD, Ma T, Thompson RC, Zhao Y, Smith L, Gasparini L, Luo Z, Xu H, Liao FF. Antidiabetic drug metformin (GlucophageR) increases biogenesis of Alzheimer's amyloid peptides via up-regulating BACE1 transcription. Proc Natl Acad Sci U S A. 2009 Mar 10;106(10):3907-12. doi: 10.1073/pnas.0807991106. Epub 2009 Feb 23. PMID 19237574
- [Background] Craft S, Raman R, Chow TW, Rafii MS, Sun CK, Rissman RA, Donohue MC, Brewer JB, Jenkins C, Harless K, Gessert D, Aisen PS. Safety, Efficacy, and Feasibility of Intranasal Insulin for the Treatment of Mild Cognitive Impairment and Alzheimer Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2020 Sep 1;77(9):1099-1109. doi: 10.1001/jamaneurol.2020.1840. PMID 32568367
- [Background] Craft S, Claxton A, Baker LD, Hanson AJ, Cholerton B, Trittschuh EH, Dahl D, Caulder E, Neth B, Montine TJ, Jung Y, Maldjian J, Whitlow C, Friedman S. Effects of Regular and Long-Acting Insulin on Cognition and Alzheimer's Disease Biomarkers: A Pilot Clinical Trial. J Alzheimers Dis. 2017;57(4):1325-1334. doi: 10.3233/JAD-161256. PMID 28372335
- [Background] Kellar D, Lockhart SN, Aisen P, Raman R, Rissman RA, Brewer J, Craft S. Intranasal Insulin Reduces White Matter Hyperintensity Progression in Association with Improvements in Cognition and CSF Biomarker Profiles in Mild Cognitive Impairment and Alzheimer's Disease. J Prev Alzheimers Dis. 2021;8(3):240-248. doi: 10.14283/jpad.2021.14. PMID 34101779
- [Background] Yoo H, Kim H, Koh I, Lee K, Ok J. Effect of Metabolic Syndrome on the Incidence of Dementia Based on National Insurance Data in Korea. Metab Syndr Relat Disord. 2022 Feb;20(1):29-35. doi: 10.1089/met.2021.0046. Epub 2021 Nov 9. PMID 34756135
- [Background] Zuin M, Roncon L, Passaro A, Cervellati C, Zuliani G. Metabolic syndrome and the risk of late onset Alzheimer's disease: An updated review and meta-analysis. Nutr Metab Cardiovasc Dis. 2021 Jul 22;31(8):2244-2252. doi: 10.1016/j.numecd.2021.03.020. Epub 2021 Apr 1. PMID 34039508
- [Background] Atti AR, Valente S, Iodice A, Caramella I, Ferrari B, Albert U, Mandelli L, De Ronchi D. Metabolic Syndrome, Mild Cognitive Impairment, and Dementia: A Meta-Analysis of Longitudinal Studies. Am J Geriatr Psychiatry. 2019 Jun;27(6):625-637. doi: 10.1016/j.jagp.2019.01.214. Epub 2019 Feb 15. PMID 30917904
- [Background] Pal K, Mukadam N, Petersen I, Cooper C. Mild cognitive impairment and progression to dementia in people with diabetes, prediabetes and metabolic syndrome: a systematic review and meta-analysis. Soc Psychiatry Psychiatr Epidemiol. 2018 Nov;53(11):1149-1160. doi: 10.1007/s00127-018-1581-3. Epub 2018 Sep 4. PMID 30182156
- [Background] Shu MJ, Zhai FF, Zhang DD, Han F, Zhou L, Ni J, Yao M, Zhang SY, Cui LY, Jin ZY, Zhu HJ, Zhu YC. Metabolic syndrome, intracranial arterial stenosis and cerebral small vessel disease in community-dwelling populations. Stroke Vasc Neurol. 2021 Dec;6(4):589-594. doi: 10.1136/svn-2020-000813. Epub 2021 Apr 26. PMID 33903177
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655
- [Background] Beeri MS, Schmeidler J, Silverman JM, Gandy S, Wysocki M, Hannigan CM, Purohit DP, Lesser G, Grossman HT, Haroutunian V. Insulin in combination with other diabetes medication is associated with less Alzheimer neuropathology. Neurology. 2008 Sep 2;71(10):750-7. doi: 10.1212/01.wnl.0000324925.95210.6d. PMID 18765651
- [Background] Katsel P, Roussos P, Beeri MS, Gama-Sosa MA, Gandy S, Khan S, Haroutunian V. Parahippocampal gyrus expression of endothelial and insulin receptor signaling pathway genes is modulated by Alzheimer's disease and normalized by treatment with anti-diabetic agents. PLoS One. 2018 Nov 1;13(11):e0206547. doi: 10.1371/journal.pone.0206547. eCollection 2018. PMID 30383799
- [Background] Doniger GM, Beeri MS, Bahar-Fuchs A, Gottlieb A, Tkachov A, Kenan H, Livny A, Bahat Y, Sharon H, Ben-Gal O, Cohen M, Zeilig G, Plotnik M. Virtual reality-based cognitive-motor training for middle-aged adults at high Alzheimer's disease risk: A randomized controlled trial. Alzheimers Dement (N Y). 2018 Mar 27;4:118-129. doi: 10.1016/j.trci.2018.02.005. eCollection 2018. PMID 29955655
- [Background] Bahar-Fuchs A, Barendse MEA, Bloom R, Ravona-Springer R, Heymann A, Dabush H, Bar L, Slater-Barkan S, Rassovsky Y, Schnaider Beeri M. Computerized Cognitive Training for Older Adults at Higher Dementia Risk due to Diabetes: Findings From a Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2020 Mar 9;75(4):747-754. doi: 10.1093/gerona/glz073. PMID 30868154
- [Background] Beeri MS, Ravona-Springer R, Moshier E, Schmeidler J, Godbold J, Karpati T, Leroith D, Koifman K, Kravitz E, Price R, Hoffman H, Silverman JM, Heymann A. The Israel Diabetes and Cognitive Decline (IDCD) study: Design and baseline characteristics. Alzheimers Dement. 2014 Nov;10(6):769-78. doi: 10.1016/j.jalz.2014.06.002. Epub 2014 Aug 20. PMID 25150735
- [Background] Ravona-Springer R, Sharvit-Ginon I, Ganmore I, Greenbaum L, Bendlin BB, Sternberg SA, Livny A, Domachevsky L, Sandler I, Ben Haim S, Golan S, Ben-Ami L, Lesman-Segev O, Manzali S, Heymann A, Beeri MS. The Israel Registry for Alzheimer's Prevention (IRAP) Study: Design and Baseline Characteristics. J Alzheimers Dis. 2020;78(2):777-788. doi: 10.3233/JAD-200623. PMID 33044181
- [Background] Hsu CL, Best JR, Davis JC, Nagamatsu LS, Wang S, Boyd LA, Hsiung GR, Voss MW, Eng JJ, Liu-Ambrose T. Aerobic exercise promotes executive functions and impacts functional neural activity among older adults with vascular cognitive impairment. Br J Sports Med. 2018 Feb;52(3):184-191. doi: 10.1136/bjsports-2016-096846. Epub 2017 Apr 21. PMID 28432077
- [Background] Morris JC, Ernesto C, Schafer K, Coats M, Leon S, Sano M, Thal LJ, Woodbury P. Clinical dementia rating training and reliability in multicenter studies: the Alzheimer's Disease Cooperative Study experience. Neurology. 1997 Jun;48(6):1508-10. doi: 10.1212/wnl.48.6.1508. PMID 9191756
- [Background] Shinar D, Gross CR, Bronstein KS, Licata-Gehr EE, Eden DT, Cabrera AR, Fishman IG, Roth AA, Barwick JA, Kunitz SC. Reliability of the activities of daily living scale and its use in telephone interview. Arch Phys Med Rehabil. 1987 Oct;68(10):723-8. PMID 3662782
- [Background] Graf C. The Lawton instrumental activities of daily living scale. Am J Nurs. 2008 Apr;108(4):52-62; quiz 62-3. doi: 10.1097/01.NAJ.0000314810.46029.74. PMID 18367931
- [Background] Birdsill AC, Carlsson CM, Willette AA, Okonkwo OC, Johnson SC, Xu G, Oh JM, Gallagher CL, Koscik RL, Jonaitis EM, Hermann BP, LaRue A, Rowley HA, Asthana S, Sager MA, Bendlin BB. Low cerebral blood flow is associated with lower memory function in metabolic syndrome. Obesity (Silver Spring). 2013 Jul;21(7):1313-20. doi: 10.1002/oby.20170. Epub 2013 May 19. PMID 23687103
- [Background] Hoscheidt SM, Kellawan JM, Berman SE, Rivera-Rivera LA, Krause RA, Oh JM, Beeri MS, Rowley HA, Wieben O, Carlsson CM, Asthana S, Johnson SC, Schrage WG, Bendlin BB. Insulin resistance is associated with lower arterial blood flow and reduced cortical perfusion in cognitively asymptomatic middle-aged adults. J Cereb Blood Flow Metab. 2017 Jun;37(6):2249-2261. doi: 10.1177/0271678X16663214. Epub 2016 Jan 1. PMID 27488909
- [Background] Merluzzi AP, Dean DC 3rd, Adluru N, Suryawanshi GS, Okonkwo OC, Oh JM, Hermann BP, Sager MA, Asthana S, Zhang H, Johnson SC, Alexander AL, Bendlin BB. Age-dependent differences in brain tissue microstructure assessed with neurite orientation dispersion and density imaging. Neurobiol Aging. 2016 Jul;43:79-88. doi: 10.1016/j.neurobiolaging.2016.03.026. Epub 2016 Apr 6. PMID 27255817
- [Background] Eren E, Hunt JFV, Shardell M, Chawla S, Tran J, Gu J, Vogt NM, Johnson SC, Bendlin BB, Kapogiannis D. Extracellular vesicle biomarkers of Alzheimer's disease associated with sub-clinical cognitive decline in late middle age. Alzheimers Dement. 2020 Sep;16(9):1293-1304. doi: 10.1002/alz.12130. Epub 2020 Jun 26. PMID 32588967
- [Background] Ashton NJ, Pascoal TA, Karikari TK, Benedet AL, Lantero-Rodriguez J, Brinkmalm G, Snellman A, Scholl M, Troakes C, Hye A, Gauthier S, Vanmechelen E, Zetterberg H, Rosa-Neto P, Blennow K. Plasma p-tau231: a new biomarker for incipient Alzheimer's disease pathology. Acta Neuropathol. 2021 May;141(5):709-724. doi: 10.1007/s00401-021-02275-6. Epub 2021 Feb 14. PMID 33585983
- [Background] Rozga M, Bittner T, Batrla R, Karl J. Preanalytical sample handling recommendations for Alzheimer's disease plasma biomarkers. Alzheimers Dement (Amst). 2019 Apr 2;11:291-300. doi: 10.1016/j.dadm.2019.02.002. eCollection 2019 Dec. PMID 30984815
- [Background] Posti JP, Takala RSK, Lagerstedt L, Dickens AM, Hossain I, Mohammadian M, Ala-Seppala H, Frantzen J, van Gils M, Hutchinson PJ, Katila AJ, Maanpaa HR, Menon DK, Newcombe VF, Tallus J, Hrusovsky K, Wilson DH, Gill J, Sanchez JC, Tenovuo O, Zetterberg H, Blennow K. Correlation of Blood Biomarkers and Biomarker Panels with Traumatic Findings on Computed Tomography after Traumatic Brain Injury. J Neurotrauma. 2019 Jul 15;36(14):2178-2189. doi: 10.1089/neu.2018.6254. Epub 2019 Apr 5. PMID 30760178
- [Background] Kellar D, Register T, Lockhart SN, Aisen P, Raman R, Rissman RA, Brewer J, Craft S. Intranasal insulin modulates cerebrospinal fluid markers of neuroinflammation in mild cognitive impairment and Alzheimer's disease: a randomized trial. Sci Rep. 2022 Jan 25;12(1):1346. doi: 10.1038/s41598-022-05165-3. PMID 35079029
- [Background] Reger MA, Watson GS, Green PS, Baker LD, Cholerton B, Fishel MA, Plymate SR, Cherrier MM, Schellenberg GD, Frey WH 2nd, Craft S. Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults. J Alzheimers Dis. 2008 Apr;13(3):323-31. doi: 10.3233/jad-2008-13309. PMID 18430999
- [Background] Smits MM, Van Raalte DH. Safety of Semaglutide. Front Endocrinol (Lausanne). 2021 Jul 7;12:645563. doi: 10.3389/fendo.2021.645563. eCollection 2021. Erratum In: Front Endocrinol (Lausanne). 2021 Nov 10;12:786732. doi: 10.3389/fendo.2021.786732. PMID 34305810
- [Background] Li A, Su X, Hu S, Wang Y. Efficacy and safety of oral semaglutide in type 2 diabetes mellitus: A systematic review and meta-analysis. Diabetes Res Clin Pract. 2023 Apr;198:110605. doi: 10.1016/j.diabres.2023.110605. Epub 2023 Mar 5. PMID 36871874
- [Background] Warren M, Chaykin L, Trachtenbarg D, Nayak G, Wijayasinghe N, Cariou B. Semaglutide as a therapeutic option for elderly patients with type 2 diabetes: Pooled analysis of the SUSTAIN 1-5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2291-2297. doi: 10.1111/dom.13331. Epub 2018 Jun 7. PMID 29687620
- [Background] Lind M, Jendle J, Torffvit O, Lager I. Glucagon-like peptide 1 (GLP-1) analogue combined with insulin reduces HbA1c and weight with low risk of hypoglycemia and high treatment satisfaction. Prim Care Diabetes. 2012 Apr;6(1):41-6. doi: 10.1016/j.pcd.2011.09.002. Epub 2011 Oct 19. PMID 22015237
- [Background] Novak V, Mantzoros CS, Novak P, McGlinchey R, Dai W, Lioutas V, Buss S, Fortier CB, Khan F, Aponte Becerra L, Ngo LH. MemAID: Memory advancement with intranasal insulin vs. placebo in type 2 diabetes and control participants: a randomized clinical trial. J Neurol. 2022 Sep;269(9):4817-4835. doi: 10.1007/s00415-022-11119-6. Epub 2022 Apr 28. PMID 35482079
- [Background] Novak P, Pimentel Maldonado DA, Novak V. Safety and preliminary efficacy of intranasal insulin for cognitive impairment in Parkinson disease and multiple system atrophy: A double-blinded placebo-controlled pilot study. PLoS One. 2019 Apr 25;14(4):e0214364. doi: 10.1371/journal.pone.0214364. eCollection 2019. PMID 31022213
- [Background] Hallschmid M, Benedict C, Schultes B, Born J, Kern W. Obese men respond to cognitive but not to catabolic brain insulin signaling. Int J Obes (Lond). 2008 Feb;32(2):275-82. doi: 10.1038/sj.ijo.0803722. Epub 2007 Sep 11. PMID 17848936
- [Background] Chang YF, Zhang D, Hu WM, Liu DX, Li L. Semaglutide-mediated protection against Abeta correlated with enhancement of autophagy and inhibition of apotosis. J Clin Neurosci. 2020 Nov;81:234-239. doi: 10.1016/j.jocn.2020.09.054. Epub 2020 Oct 14. PMID 33222922
- [Background] During MJ, Cao L, Zuzga DS, Francis JS, Fitzsimons HL, Jiao X, Bland RJ, Klugmann M, Banks WA, Drucker DJ, Haile CN. Glucagon-like peptide-1 receptor is involved in learning and neuroprotection. Nat Med. 2003 Sep;9(9):1173-9. doi: 10.1038/nm919. Epub 2003 Aug 17. PMID 12925848
- [Background] Goke R, Larsen PJ, Mikkelsen JD, Sheikh SP. Distribution of GLP-1 binding sites in the rat brain: evidence that exendin-4 is a ligand of brain GLP-1 binding sites. Eur J Neurosci. 1995 Nov 1;7(11):2294-300. doi: 10.1111/j.1460-9568.1995.tb00650.x. PMID 8563978
- [Background] Femminella GD, Frangou E, Love SB, Busza G, Holmes C, Ritchie C, Lawrence R, McFarlane B, Tadros G, Ridha BH, Bannister C, Walker Z, Archer H, Coulthard E, Underwood BR, Prasanna A, Koranteng P, Karim S, Junaid K, McGuinness B, Nilforooshan R, Macharouthu A, Donaldson A, Thacker S, Russell G, Malik N, Mate V, Knight L, Kshemendran S, Harrison J, Holscher C, Brooks DJ, Passmore AP, Ballard C, Edison P. Evaluating the effects of the novel GLP-1 analogue liraglutide in Alzheimer's disease: study protocol for a randomised controlled trial (ELAD study). Trials. 2019 Apr 3;20(1):191. doi: 10.1186/s13063-019-3259-x. Erratum In: Trials. 2020 Jul 19;21(1):660. doi: 10.1186/s13063-020-04608-4. PMID 30944040
- [Background] Robinson A, Lubitz I, Atrakchi-Baranes D, Licht-Murava A, Katsel P, Leroith D, Liraz-Zaltsman S, Haroutunian V, Beeri MS. Combination of Insulin with a GLP1 Agonist Is Associated with Better Memory and Normal Expression of Insulin Receptor Pathway Genes in a Mouse Model of Alzheimer's Disease. J Mol Neurosci. 2019 Apr;67(4):504-510. doi: 10.1007/s12031-019-1257-9. Epub 2019 Jan 11. PMID 30635783
- [Background] Avgerinos KI, Ferrucci L, Kapogiannis D. Effects of monoclonal antibodies against amyloid-beta on clinical and biomarker outcomes and adverse event risks: A systematic review and meta-analysis of phase III RCTs in Alzheimer's disease. Ageing Res Rev. 2021 Jul;68:101339. doi: 10.1016/j.arr.2021.101339. Epub 2021 Apr 5. PMID 33831607
- [Background] Cho Y, Han K, Kim DH, Park YM, Yoon KH, Kim MK, Lee SH. Cumulative Exposure to Metabolic Syndrome Components and the Risk of Dementia: A Nationwide Population-Based Study. Endocrinol Metab (Seoul). 2021 Apr;36(2):424-435. doi: 10.3803/EnM.2020.935. Epub 2021 Apr 14. PMID 33849249
- [Background] Gaubert M, Lange C, Garnier-Crussard A, Kobe T, Bougacha S, Gonneaud J, de Flores R, Tomadesso C, Mezenge F, Landeau B, de la Sayette V, Chetelat G, Wirth M. Topographic patterns of white matter hyperintensities are associated with multimodal neuroimaging biomarkers of Alzheimer's disease. Alzheimers Res Ther. 2021 Jan 18;13(1):29. doi: 10.1186/s13195-020-00759-3. PMID 33461618
- [Background] Heiss WD. The Additional Value of PET in the Assessment of Cerebral Small Vessel Disease. J Nucl Med. 2018 Nov;59(11):1660-1664. doi: 10.2967/jnumed.118.214270. Epub 2018 Jun 29. PMID 29959217
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Petersen RC, Weiner MW, Aisen PS, Shaw LM, Vemuri P, Wiste HJ, Weigand SD, Lesnick TG, Pankratz VS, Donohue MC, Trojanowski JQ. Tracking pathophysiological processes in Alzheimer's disease: an updated hypothetical model of dynamic biomarkers. Lancet Neurol. 2013 Feb;12(2):207-16. doi: 10.1016/S1474-4422(12)70291-0. PMID 23332364
- [Background] Qiu M, Ding LL, Zhang M, Zhou HR. Safety of four SGLT2 inhibitors in three chronic diseases: A meta-analysis of large randomized trials of SGLT2 inhibitors. Diab Vasc Dis Res. 2021 Mar-Apr;18(2):14791641211011016. doi: 10.1177/14791641211011016. PMID 33887983
- [Background] Douros A, Lix LM, Fralick M, Dell'Aniello S, Shah BR, Ronksley PE, Tremblay E, Hu N, Alessi-Severini S, Fisher A, Bugden SC, Ernst P, Filion KB; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Sodium-Glucose Cotransporter-2 Inhibitors and the Risk for Diabetic Ketoacidosis : A Multicenter Cohort Study. Ann Intern Med. 2020 Sep 15;173(6):417-425. doi: 10.7326/M20-0289. Epub 2020 Jul 28. PMID 32716707
- [Background] Seidu S, Kunutsor SK, Topsever P, Khunti K. Benefits and harms of sodium-glucose co-transporter-2 inhibitors (SGLT2-I) and renin-angiotensin-aldosterone system inhibitors (RAAS-I) versus SGLT2-Is alone in patients with type 2 diabetes: A systematic review and meta-analysis of randomized controlled trials. Endocrinol Diabetes Metab. 2022 Jan;5(1):e00303. doi: 10.1002/edm2.303. Epub 2021 Oct 12. PMID 34636161
- [Background] Heymann AD, Chodick G, Halkin H, Karasik A, Shalev V, Shemer J, Kokia E. The implementation of managed care for diabetes using medical informatics in a large Preferred Provider Organization. Diabetes Res Clin Pract. 2006 Mar;71(3):290-8. doi: 10.1016/j.diabres.2005.07.002. Epub 2005 Aug 19. PMID 16112245
- [Background] BenAri O, Efrati S, Sano M, Bendlin BB, Lin H, Liu X, Sela I, Almog G, Livny A, Sandler I, Ben-Haim S, Sagi R, LeRoith D, Schnaider Beeri M, Ravona-Springer R. A double-blind placebo-controlled clinical trial testing the effect of hyperbaric oxygen therapy on brain and cognitive outcomes of mildly cognitively impaired elderly with type 2 diabetes: Study design. Alzheimers Dement (N Y). 2020 Apr 13;6(1):e12008. doi: 10.1002/trc2.12008. eCollection 2020. PMID 32296731